CLINICAL TRIAL: NCT02638142
Title: Continuous Versus Bolus Intermittent Loop Diuretic Infusion in Acutely Decompensated Heart Failure: Evaluation of Renal Function, Congestion Signs, BNP and Outcome
Brief Title: Loop Diuretic Therapy in Acutely Decompensated Heart Failure
Acronym: DIUR-AHF
Status: Recruiting | Type: Observational
Sponsor: University of Siena (Other)
Collaborators: University of Roma La Sapienza (Other); Ospedale Regina Montis Regalis (Other); University of Naples (Other); A.O.U. Città della Salute e della Scienza (Other); University of Milan (Other)
Responsible Party: Principal Investigator, Alberto Palazzuoli MD PhD, Medical Doctor, Cardiologist, University of Siena
Other Study IDs: DIUR-AHF
Record Dates: First submitted 2015-12-09; First posted 2015-12-22 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Heart Failure
Keywords: loop diuretic; heart failure; renal dysfunction; congestion signs; BNP
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Continuous Furosemide Infusion: continuous intravenous furosemide infusion
  Interventions: Drug: Continuous Furosemide Infusion
- Intermittent Furosemide Infusion: bolus intermittent intravenous furosemide infusion
  Interventions: Drug: Intermittent Furosemide Infusion

INTERVENTIONS:
Drug: Continuous Furosemide Infusion — Intravenous continuous Furosemide infusion
  Other Names: cIV
  Groups: Continuous Furosemide Infusion
Drug: Intermittent Furosemide Infusion — Intravenous bolus intermittent Furosemide Infusion
  Other Names: iIV
  Groups: Intermittent Furosemide Infusion

SUMMARY:
DiurHF is a prospective, multicenter, observational, study that compares continuous with intermittent infusion of furosemide in patients admitted with a diagnosis of ADHF. Previous pilot study design was planned to anticipate a larger multicenter trial able to definitively evaluate the optimal loop diuretic use strategy in patients with ADHF.

DETAILED DESCRIPTION:
The use of intravenous loop diuretics is a cornerstone of therapy for acutely decompensated heart failure (ADHF); significant concerns have been raised regarding risks and benefits of loop diuretics, particularly about dosage and administration regimen.

Recent guidelines recommend the use of these drugs to reduce left ventricular filling pressure, avoid pulmonary edema, and alleviate peripheral fluid retention.

Some studies have provided guidelines for the administration of these drugs in clinical practice, but data interpretation remains challenging due to the frequent exclusion of patients with kidney disease from major ADHF clinical trials. Therefore, it is not clear if continuous infusion is better than intermittent boluses in terms of decongestion, maintenance of renal filtration function and prognosis.

On the other hand, continuous administration should provide a more constant delivery of the drug into the tubule, potentially reducing these phenomena.

The aim of the study is to evaluate the better loop diuretic intravenous administration in terms of renal function, congestion signs, BNP and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years;
* Patients with diagnosis of ADHF(dyspnea, orthopnea, peripheral edema or major fatigue and at least two clinical signs including rales, hepatomegaly, pulmonary congestion on chest radiography, jugular vein dilatation, or a third heart sound);
* Blood BNP > 100 pg/mL;

ADHF: Acute Decompensated Heart Failure; BNP: B-type Natriuretic Peptide; IV: IntraVenous; LVEF: Left Ventricular Ejection Fraction.

Exclusion Criteria:

* Patients who receive more than 40 mg of IV furosemide;
* End-Stage renal disease or renal replacement therapy;
* Recent myocardial infarction (within thirty days of screening);
* Systolic blood pressure < 80 mmHg;
* Creatinine levels > 4 mg/dL;
* Patients affected by sepsis, liver diseases, inflammatory diseases or neoplastic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who met diagnostic criteria for ADHF, independently from systolic function by exhibiting: at least one symptom at rest between dyspnea, orthopnea, peripheral edema and major fatigue; and at least two clinical signs including rales, pulmonary congestion on chest radiography, jugular vein dilatation and a third heart sound. An elevation in blood BNP >100 pg/ml was considered supportive for a diagnosis of ADHF
Sampling Method: Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac death and rehospitalization for HF | 180 days
  Number of participant who are affected by cardiovascular death or rehospitalization within 180 days from discharge.

SECONDARY OUTCOMES:
length of hospital stay (days) | From date of randomization until the discharge (7-12 days)
  evaluation of length of hospital stay (days) in the two groups
Inotropes agents | From date of randomization until the discharge (7-12 days)
  Need to use inotropes agents during the treatment
hypertonic saline solution | From date of randomization until the discharge (7-12 days)
  need to use hypertonic saline solution during the treatment
Acute kidney injury | From date of randomization until the discharge (7-12 days)
  changes of renal function in terms of creatinine and estimated glomerular filtration rate (eGFR) comparing continuous vs intermittent administration
Body weight changes | from admission to discharge (7-12 days)
  Body weight changes in two groups from the admission to discharge
Diuresis | from admission to discharge (7-12 days)
  mean urine output in two groups from the admission to discharge
BNP changes | From date of randomization until the discharge (7-12 days)
  mean paired changes of B-type natriuretic peptide (BNP) in the two groups during hospitalization.
BUN changes | From date of randomization until the discharge (7-12 days)
  mean paired changes of blood urea nitrogen (BUN) in the two groups during hospitalization.
Reduction of edema | From date of randomization until the discharge (7-12 days)
  Evaluation of edema regression (or not) after treatment in the two groups.
Reduction of dyspnea | From date of randomization until the discharge (7-12 days)
  Evaluation of dyspnea scale reduction (or not) after treatment in the two groups.
Regression of pulmonary congestion | From date of randomization
  Evaluation of pulmonary congestion regression (or not) after treatment in the two groups, considering Chest X-ray at admission and at discharge
Diuretic efficiency: (Weight loss/days of infusion)/ (Mean daily furosemide dosage/40 mg of furosemide) | From hospital admission until the discharge (7-12 days)
  Evaluation of persistence of congestion (or not) and incidence of AKI (or not) according to quartiles of diuretic efficiency.
High (> 125 mg/die) versus low (<125 mg/die) intravenous diuretic dosage | 180 days
  Number of patients with high in-hospital diuretic dosage who were affected by adverse outcome.
Diuretic efficiency: (Weight loss/days of infusion)/ (Mean daily furosemide dosage/40 mg of furosemide) | 180 days
  Number of patients (according quartiles of diuretic efficiency) who were affected by adverse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Palazzuoli, MD, Principal Investigator — University of Siena
Locations (4):
- Italy (4):
  - Ospedale Madonna della Navicella, Chioggia, Venezia
  - Azienda Ospedaliera di Padova, Padua
  - University of Rome La Sapienza, Roma
  - Department of Internal Medicine, Cardiovascular Diseases Unit, Siena

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Palazzuoli A, Pellegrini M, Ruocco G, Martini G, Franci B, Campagna MS, Gilleman M, Nuti R, McCullough PA, Ronco C. Continuous versus bolus intermittent loop diuretic infusion in acutely decompensated heart failure: a prospective randomized trial. Crit Care. 2014 Jun 28;18(3):R134. doi: 10.1186/cc13952. PMID 24974232
- [Result] Felker GM, Lee KL, Bull DA, Redfield MM, Stevenson LW, Goldsmith SR, LeWinter MM, Deswal A, Rouleau JL, Ofili EO, Anstrom KJ, Hernandez AF, McNulty SE, Velazquez EJ, Kfoury AG, Chen HH, Givertz MM, Semigran MJ, Bart BA, Mascette AM, Braunwald E, O'Connor CM; NHLBI Heart Failure Clinical Research Network. Diuretic strategies in patients with acute decompensated heart failure. N Engl J Med. 2011 Mar 3;364(9):797-805. doi: 10.1056/NEJMoa1005419. PMID 21366472
- [Result] Lala A, McNulty SE, Mentz RJ, Dunlay SM, Vader JM, AbouEzzeddine OF, DeVore AD, Khazanie P, Redfield MM, Goldsmith SR, Bart BA, Anstrom KJ, Felker GM, Hernandez AF, Stevenson LW. Relief and Recurrence of Congestion During and After Hospitalization for Acute Heart Failure: Insights From Diuretic Optimization Strategy Evaluation in Acute Decompensated Heart Failure (DOSE-AHF) and Cardiorenal Rescue Study in Acute Decompensated Heart Failure (CARESS-HF). Circ Heart Fail. 2015 Jul;8(4):741-8. doi: 10.1161/CIRCHEARTFAILURE.114.001957. Epub 2015 Jun 3. PMID 26041600
- [Result] ter Maaten JM, Dunning AM, Valente MA, Damman K, Ezekowitz JA, Califf RM, Starling RC, van der Meer P, O'Connor CM, Schulte PJ, Testani JM, Hernandez AF, Tang WH, Voors AA. Diuretic response in acute heart failure-an analysis from ASCEND-HF. Am Heart J. 2015 Aug;170(2):313-21. doi: 10.1016/j.ahj.2015.05.003. Epub 2015 May 9. PMID 26299229
- [Result] Voors AA, Davison BA, Teerlink JR, Felker GM, Cotter G, Filippatos G, Greenberg BH, Pang PS, Levin B, Hua TA, Severin T, Ponikowski P, Metra M; RELAX-AHF Investigators. Diuretic response in patients with acute decompensated heart failure: characteristics and clinical outcome--an analysis from RELAX-AHF. Eur J Heart Fail. 2014 Nov;16(11):1230-40. doi: 10.1002/ejhf.170. Epub 2014 Oct 7. PMID 25287144
- [Derived] Palazzuoli A, Dini FL, Pugliese NR, Ruocco G, Severino P, Vizza D, Carbonara R, Passantino A, Carluccio E. Right Ventricular-Pulmonary Artery Uncoupling and Strain in Acute Heart Failure. J Am Heart Assoc. 2025 May 6;14(9):e039858. doi: 10.1161/JAHA.124.039858. Epub 2025 May 2. PMID 40314350
- [Derived] Palazzuoli A, Ruocco G, Vescovo G, Valle R, Di Somma S, Nuti R. Rationale and study design of intravenous loop diuretic administration in acute heart failure: DIUR-AHF. ESC Heart Fail. 2017 Nov;4(4):479-486. doi: 10.1002/ehf2.12226. Epub 2017 Oct 4. PMID 28980452